CLINICAL TRIAL: NCT02488655
Title: Treatment of Breast Fibroadenoma With FastScan High Intensity Focused Ultrasound (HIFU)
Brief Title: Treatment of Breast Fibroadenoma With FastScan HIFU
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Theraclion (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HIFU/BG/FA/FS/2015
Record Dates: First submitted 2015-06-24; First posted 2015-07-02 (Estimated); Last update posted 2021-10-19 (Actual); Status verified 2021-10

CONDITIONS: Breast Fibroadenoma
MeSH Terms: conditions — Fibroadenoma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Echopulse (Experimental): Echopulse HIFU
  Interventions: Device: Echopulse

INTERVENTIONS:
Device: Echopulse — HIFU Under ultrasound guidance
  Other Names: Echopulse HIFU

SUMMARY:
This study evaluates the efficacy of the HIFU for the treatment of breast fibroadenoma with the FastScan version using assessment of patient experience and adverse event reporting.

DETAILED DESCRIPTION:
Echopulse is specially designed, manufactured and CE marked for treating breast fibroadenoma. HIFU is a completely alternative to surgery which utilizes high-energy ultrasound to deliver a large amount of sound energy to a focal point to rapidly induce tissue heating to 85-90°C.This initiates tissue coagulation followed by tissue necrosis ablating the targeted area.

In a previous european feasibility study performed at 4 sites (France and Bulgaria), 51 fibroadenomas in 42 patients were treated. The HIFU treatment was well tolerated and showed efficacy (mean volume reduction of 72.5% +/-16.7 at 12 months follow-up.

ELIGIBILITY:
Inclusion Criteria:

* Female patients 18 years or older with one diagnosed breast fibroadenoma.
* Diagnosis of fibroadenoma must be based on :

  * clinical examination,
  * ultrasound image alone for patients under 35 years old. For women older than 35 years, a mammogram will be performed in addition to ultrasound. The BI-RADS (Breast Imaging, Reporting and Data System) score of this mammogram must be less than 3.
  * histologic confirmation after core needle biopsy by two independent readers (biopsy must be performed at least two weeks before therapy unless a microbiopsy has been already done less than 3 months before inclusion visit and histopathology slices are available).
* The requirements for the distance from the skin and the following regions of the fibroadenoma are:

  * ≤ 23 mm from the posterior border of the fibroadenoma
  * ≥ 5 mm from the anterior border of the fibroadenoma
  * ≥ 11mm from the focal point of the HIFU treatment. These criteria shall be evaluated immediately prior to treatment once breast is immobilized and potentially compressed
* The rib cage should not be in the prefocal ultrasound path or behind the target fibroadenoma (minimum distance behind the focal point= 10 mm). This criterion shall only be reached in treatment conditions, once breast is immobilized and potentially compressed.
* Patient's fibroadenoma is 1 cm or greater at its largest dimension
* Fibroadenoma is palpable
* Patient has signed a written informed consent.

Exclusion Criteria:

* Patient who is pregnant or lactating.
* Patient with a BI-RADS score > 2 at the mammogram, or presence of microcalcifications within the lesion.
* Patient with history of breast cancer or history
* Patient with history of laser or radiation therapy to the target breast
* Patient with breast implants in the target breast
* Patient with a breast cyst
* Patient's fibroadenoma not clearly visible on the ultrasound images (in B mode) at the inclusion visit
* Patient participating in other trials using drugs or devices.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2015-06; Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
Number of participants with adverse events | 1 day post treatment
Number of participants with adverse events | 3 days post treatment
Number of participants with adverse events | 7 days post treatment
Change from Baseline volume of the fibroadenoma at 6 months | 6 months post treament
Change from Baseline Patient pain intensity score (100mm visual analog scale) at 1 day | 1 day post treatment
Change from Baseline Patient pain intensity score (100mm visual analog scale) at 3 days | 3 days post treatment
Change from Baseline Patient pain intensity score (100mm visual analog scale) at 7 days | 7 days post treatment
Patient satisfaction questionnaire | 6 months post treatment

SECONDARY OUTCOMES:
Number of participants with absence of palpable lesion | 3 months post treatment
Number of participants with absence of palpable lesion | 6 months post treatment
Patient Cosmetic evaluation as measured by questionnaire | 6 months post treatment
Investigator rated evaluation of the device | Post treatment Day 0
Change from Baseline gland vascularization at 3 months | 3 months post treatment
Change from Baseline gland vascularization at 6 months | 6 months post treatment

CONTACTS AND LOCATIONS:
Overall Officials: Roussanka Kovatcheva, Prof., Principal Investigator — roussanka_kov@yahoo.com
Locations (1):
- University Hospital of Endocrinology USBALE, Sofia, Bulgaria